CLINICAL TRIAL: NCT06217445
Title: Effect of High Intensity Focused Ultrasound on Sleep Quality Measures in Obese Doubled Chin Women
Brief Title: Effect of HIFU on Sleep Quality Measures in Obese Doubled Chin Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Tharwat Mousa Ahmed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIFU treatment on obese women
Record Dates: First submitted 2024-01-06; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: OBESITY
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: parallel study is type of clinical study in which two or more groups of participants receive different interventions.
Who Masked: Participant, Outcomes Assessor
Masking Description: DOUBLE BLIND
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU plus exercises (Experimental): 1. A physician or technician first cleans the target area.
  2. They may apply a topical anesthetic cream before starting.
  3. The physician or technician then applies an ultrasound gel.
  4. The HIFU device is placed against the skin.
  5. Using an ultrasound viewer, the physician or technician adjusts the device to the right setting.
  6. Ultrasound energy is then delivered to the target area in short pulses for roughly 30 to 90 minutes.
  7. The device is removed.
  Interventions: Device: high intensity focused ultrasound
- doubled chin exercises (Experimental): 1. Straight jaw jut
  2. Ball exercise
  3. Pucker up
     .
  4. Tongue stretch
  5. Neck stretch
  6. Bottom jaw jut
  Interventions: Other: Doubled chin exercises

INTERVENTIONS:
Device: high intensity focused ultrasound — High-intensity focused ultrasound (HIFU) therapy is becoming more familiar in medical field because it is non-invasive technique with fewer side effects and provides promising therapeutic results. Several HIFU therapy applications have approved by many approval authorities of deferent countries since last decade
  Arms: HIFU plus exercises
Other: Doubled chin exercises — 1. Straight jaw jut. 2-ball exercise. 3-Pucker up 4. Tongue stretch 5. Neck stretch 6-bottom jaw jut.
  Arms: doubled chin exercises

SUMMARY:
This study will be conducted to demonstrate any effect of high intensity focused ultrasound on sleep quality measures in obese doubled chin women.

DETAILED DESCRIPTION:
PURPOSE:

This study will be conducted to demonstrate any effect of high intensity focused ultrasound on sleep quality measures in obese doubled chin women.

BACKGROUND:

High-intensity focused ultrasound (HIFU) therapy is becoming more familiar in medical field because it is non-invasive technique with fewer side effects and provides promising therapeutic results. Several HIFU therapy applications have approved by many approval authorities of deferent countries since last decade.

HIFU cauterizes tissue from outside the body by focusing ultrasonic waves from a transducer with many ultrasonic sources on a single point, known as the target tumor .This modality is groundbreaking because it only causes coagulative necrosis via thermal and non-thermal energy (mainly cavitation) to the focal area, with hardly any impact on the intervening tissue outside the focal area.

Central obesity is significant predictor of metabolic syndrome and is associated with an increased risk of many medical conditions, including cardiovascular diseases (CVD), stroke , type 2 diabetes mellitus, hypertension , various types of cancer (e.g. colorectum, pancreas, endometrium, and breast) and all-cause mortality

Hypotheses of the study(Null) There is no significant effect of High Intensity Focused Ultrasound on sleep quality measures in obese doubled chin women.

Statement of the problem:

Is there any effect of high intensity focused ultrasound on sleep quality measures in obese doubled chin women?

ELIGIBILITY:
Inclusion Criteria:

* All patients that will be included in this study will meet the following criteria:

  1. Female subjects with age ranged from 35 to 50 years old.
  2. BMI will be 30-39.9. Class I,II

BMI was classified into six groups:

underweight (<18.5 kg/m2) normal (18.5-24.9 kg/m2) pre-obesity (25-29.9 kg/m2) obesity class I (30-34.9 kg/m2) obesity class II (35-39.9 kg/m2) obesity class III (>40 kg/m2) 3. Clinically and medically stable. 4. Able to understand the requirements of the study. 5.Thyroxin normal level( thyroid-stimulating hormone) (0.35 and 5.0milli-International unit( mIU/L)

Exclusion Criteria:

- The potential participants will be excluded if they meet one of the following criteria:

1. Neurological conditions (e.g., stroke history, Parkinson's disease).
2. Presence of an acute illness.
3. Renal and Hepatic diseases.
4. Patient undergoes chemotherapy.
5. Recent surgery.
6. Any contraindications for using HIFU such as:pregnancy ,metal prosthesis or implants,epilepsy,diabetes, autoimmune conditions,heart diseases including pacemaker,thrombosis .

8-BMI less than 30 and more than 39.9. 9-Age less than 35 and more than 50. 10-Male subjects.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-04-06 (Estimated); Study Completion 2024-04-06 (Estimated)

PRIMARY OUTCOMES:
submental fat scale | 3 months
  It ranges from 0 (no localised sub-mental fat) to 4 (extreme submental convexity). The ideal patient for would be someone who is a '2' or '3' on sub-mental scale, so someone with moderate to severe sub-mental fullness
Spirometric assessment for obesity | 3 months
  patients underwent spirometry tests with measurement of forced expiratory volume in first second (FEV1), forced vital capacity (FVC)and(MVV)
Impact of Weight on Quality of Life Assessment Tools: | 3 months
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated, 31-item, self-report measure of obesity-specific quality of life in adults, available in multiple languages. scale structure of the IWQOL-Lite has been verified with confirmatory factor analysis, and IWQOL-Lite scores are sensitive to changes in weight. There is strong evidence for validity and reliability.
  ▪ In addition to a total score, there are scores on five domains:
  * Physical function (11 items)
  * Self-esteem (7 items)
  * Sexual life (4 items)
  * Public distress (5 items)
  * Work (4 items) Scores range from 0 to 100, with 100 representing the best quality of life. Raw scores are no longer used for reporting

SECONDARY OUTCOMES:
Assessment of hormonal changes | 3 months
  there might also be deposits of fat around the neck, resulting in a double chin or moon face appearance. This appearance has been linked to glucose and cortisol imbalances, and diminished thyroid function. SO measure cortisol hormone.
  A cortisol test often uses a sample of blood drawn at a lab. cortisol level is a blood test that measures the amount of cortisol, a steroid hormone produced by the adrenal cortex.
  Normal values for a blood sample taken at 8 in the morning are 5 to 25 mcg/dL.
  A higher than normal level may indicate:
  Cushing disease Ectopic Cushing syndrome, in which a tumor outside the pituitary or adrenal glands makes too much ACTH Tumor of the adrenal gland,stress,acute illness
  A lower than normal level may indicate:
  Addison disease Suppression of normal pituitary or adrenal function by glucocorticoid medicines
Assessment of snoring | 3 months
  scale from 0-5 . 0 indicate no snoring. 1 indicate rarely slight snoring depends on sleep position. 2 indicate continuous slight snoring without hypopnea or apnea. 3 indicate sometimes loud snoring without hypopnea or apnea. 4 indicate continuous loud snoring without hypopnea or apnea.5 indicate continuous loud snoring with hypopnea or apnea
Assessment of sleep apnea: | 3 months
  The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep.
  The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. The AHI values for adults are categorized as:
  * Normal: AHI<5
  * Mild sleep apnea: 5≤AHI<15
  * Moderate sleep apnea: 15≤AHI<30
  * Severe sleep apnea: AHI≥30

CONTACTS AND LOCATIONS:
Overall Officials: HANI EZZAT OBAYA, prof ass.dr, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

REFERENCES:
- [Background] Ayatollahi A, Gholami J, Saberi M, Hosseini H, Firooz A. Systematic review and meta-analysis of safety and efficacy of high-intensity focused ultrasound (HIFU) for face and neck rejuvenation. Lasers Med Sci. 2020 Jul;35(5):1007-1024. doi: 10.1007/s10103-020-02957-9. Epub 2020 Feb 5. PMID 32026164
- [Background] Zhou X, Li Y, Zhu Q, Luo J, Cao L, Quetai J, Li F, Tang MX, Wang Z. A Theragnostic HIFU Transducer and System for Inherently Registered Imaging and Therapy. IEEE Trans Biomed Eng. 2023 Dec;70(12):3413-3424. doi: 10.1109/TBME.2023.3287870. Epub 2023 Nov 21. PMID 37339046